CLINICAL TRIAL: NCT03178838
Title: Preliminary Clinical Study of the Presence of Trichomonas Tenax and Entamoeba Gingivalis in Patients With Periodontitis Consulting to CHU of Nancy, in Periodontal Department.
Brief Title: Clinical Study of the Presence of Trichomonas Tenax and Entamoeba Gingivalis in Patients With Periodontitis
Acronym: Paro-Proto 2
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/PARO-PROTO-BISSON/VS
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The buccal cavity presents microorganismes whose the number and composition vary with oral hygiene and medical context (pathologies and associated drug therapies) of the patient. More than 1200 bacterial species have been identified, and among them, 400 are inhabitants of the sub-gingival biofilm. Among all these microorganismes, only 20 species participate to the etiopathogenesis of periodontal diseases.Some are recognised as major periodontopathogens other play unclear role in this pathology. They belong respectively to the red and orange complex of Socransky et al. (1998).

Other microorganismes such as virures, yeasts and protozoans could potentially impact the emergence and development of periodontal diseases. The presence of protozoans in periodontitis have been investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years-old
* Consulting in periodontal department of CHU, Nancy
* Patient with moderate to severe periodontitis
* At least 2 periodontal sites with PPD≥ 4mm and One healthy site
* No scaling root planning in the last 6 months
* Patients insured under the French social security system

Exclusion Criteria:

* Pregnant patients
* Patients with antibiotic therapy, and/or all medecines which could modify the buccal microbiota in the last 6 months
* Tooth with endodontic periapical lesion
* Patients having a scaling root planning in the last 6 months
* Patient with guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in the periodontal department of CHU, Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2014-11-11 (Actual); Study Completion 2014-11-11 (Actual)

PRIMARY OUTCOMES:
Presence of protozoans | baseline

SECONDARY OUTCOMES:
Periodontal pocket depth (mm) | baseline
Clinical attachment loss (mm) | baseline
Plaque and gingival index | baseline
Mobility of the tooth (Yes/No) | baseline
Presence of bleeding on probing (Yes/No) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BISSON, PhD, Principal Investigator — CHRU Nancy / Université de Lorraine

IPD SHARING:
Plan to Share IPD: No
Commission Nationale de l'Informatique et des libertés